CLINICAL TRIAL: NCT02965235
Title: Correlations of Epigenetic Changes With POCD in Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Ru-Ping Dai, Professor, MD, PhD, Central South University
Other Study IDs: XYEYYLH20151209
Record Dates: First submitted 2016-11-14; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For analysis of epigenetic changes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non-POCD: Patients who don't develop POCD after surgery.
- POCD: Patients who develop POCD after surgery.

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a subtle cognitive dysfunction, especially postoperative memory impairment lasting for weeks or months. The underlying pathophysiological mechanism of POCD remain unclear. The aim of this study is to explore the epigenetic changes during perioperative period and its correlation with POCD in surgical patients.

DETAILED DESCRIPTION:
The incidence of postoperative cognitive dysfunction (POCD) in elderly patients ranges widely from 16% to 21% and is associated with adverse outcomes. The exact cause of POCD remains unknown. Extensive studies report that epigenetic modification, including the alteration of DNA methylation and chromatin structure, plays an important part in the regulation of memory and learning. The present study thus hypothesize that epigenetic modification may increase the risk for POCD. The present study will enrolled the elderly patients (aged≥65) and young and middle-aged patents (aged 20-50) who are planning to undergo elective noncardiac surgery under general anesthesia. Perioperative clinical characteristics of all patients will be recorded. Participants enrolled will be evaluated for POCD with Mini-Mental State Examination (MMSE) on preoperative day, postoperative days 1. Postoperative pain will be evaluated by the numerical rating scale (NRS). The patients' blood will be collected in the morning on the day before surgery and after surgery when they recover consciousness for the detection of concentration of 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) by enzyme-linked immunosorbent assays (ELISA).

The present study may help to find whether epigenetic changes will occur after surgical and anesthesia stress and will be an important factor for POCD in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

•ASA Grade I to III Age >65 BMI 18-28kg/m2 Patients undergoing abdominal surgery,orthopedic surgery and spinal surgery

Exclusion Criteria:

* Exclusion Criteria:

  * do not consent, Patients with mini mental state examination (MMSE)score of ≤20 at screening severe heart,kidney or lung disfunction;unstable angina undergoing abdominal operation previously refuse to use PCA unexpected surgical complication such as bleeding; psychiatric disorders; drug or alcohol abuse

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: central south university,xiangya 2nd hospital,general surgery department
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of epigenetic changes with POCD | 24 hours
  The present study will examine concentration of 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) in whole blood by enzyme-linked immunosorbent assays (ELISA) to determine the correlation of epigenetic changes with POCD in surgical patients.

SECONDARY OUTCOMES:
The effects of surgical and anesthesia stress on epigenetic changes | 24 hours
  Numerous studies have reported that both acute and chronic stress can cause epigenetic modification. Surgical stress also belongs to acute stress during perioperative period. Thus the present study will compare concentration of 5-methylcytosine (5mC) and 5-hydroxymethylcytosine (5hmC) before and after operation to determine whether surgical and anesthesia stress will induce epigenetic changes.

CONTACTS AND LOCATIONS:
Overall Officials: Ruping Dai, MD, Principal Investigator — The Second Xiangya Hospital, Central South University
Locations (1):
- Department of Anesthesiology, The Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Wu TT, Tang L, Liu Q, Mao XZ, Xu JM, Dai RP. Association of global DNA hypomethylation with post-operative cognitive dysfunction in elderly patients undergoing hip surgery. Acta Anaesthesiol Scand. 2020 Mar;64(3):354-360. doi: 10.1111/aas.13502. Epub 2019 Nov 23. PMID 31715023